CLINICAL TRIAL: NCT03057158
Title: Epigenomics in Insulin Resistance Associated Overactive Bladder.
Brief Title: Genomics and Epigenomics for New Insights in fEmale OAB (GENIE) Study
Acronym: GENIE
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00079255; 302-0870 (Other Grant/Funding Number: NIDDK)
Record Dates: First submitted 2017-02-13; First posted 2017-02-17 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2019-11

CONDITIONS: Overactive Bladder; Insulin Resistance
Keywords: OAB; Insulin resistance; diabetes; pre-diabetes
MeSH Terms: conditions — Urinary Bladder, Overactive; Insulin Resistance; Diabetes Mellitus; Glucose Intolerance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine and blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1: Women with Urgency Incontinence (At least three times per week) greater than three months, and without insulin resistance.
- 2: Women with insulin resistance (pre-diabetes or diabetes based on Hemoglobin A1C).
- 3: Women with both UUI (at least three times per week for over three months) and Insulin Resistance (pre-diabetes or diabetes based on Hemoglobin A1C).
- 4: Healthy Volunteers

SUMMARY:
Millions of women suffer from overactive bladder, and the changes in bladder function affect their quality of life. The study team believes that it needs to be better understand why women get overactive bladder in the first place so that better treatments can eventually be offered.

The purpose of this study is to determine why women with insulin resistance are more likely to get overactive bladder. Overactive bladder is a type of bladder control problem that can cause some women to have bladder leakage. This problem is more common in women with diabetes and pre-diabetes, but it isn't known why.

DETAILED DESCRIPTION:
The methylation of cytosines in CpG sites can have profound effects on the ability of genes to be transcribed. To clarify and distinguish the specific methylation changes responsible for overactive bladder (OAB) in those with insulin resistance (IR), the investigator will compare three well-characterized groups of women: 1) OAB and IR; 2) IR only (no OAB); and 3) OAB only (no IR). In this proposal the investigator is only studying women since they are more likely to be affected by OAB with incontinence, the investigator wants to study pure cohorts of patients, and because this is the clinical population cared for by the primary investigator. The plan for future investigations is to apply these findings to broader groups to better understand gender and racial differences.

In Specific Aim 1, the investigator will conduct an epigenome-wide association study (EWAS) study, followed by targeted validation studies to determine whether CpG sites throughout the genome are differentially methylated in well-characterized and matched cohorts, while controlling for the effects of insulin-resistance. In Specific Aim 2, the investigator will assess for differential expression of candidate loci in relation to methylation. RNA-sequencing (RNA-seq) will be used to establish differences in the transcriptome between extreme phenotypes of OAB+IR and OAB alone. The investigator will then use quantitative polymerase chain reaction (qPCR) to validate expression differences in all cohorts, and to confirm differences in candidate loci that are confirmed in experiments from Aim 1. The investigator will proceed with bioinformatic pathway analyses to identify the function and interdependence of genes with altered expression and altered methylation profiles. In Specific Aim 3, the investigator will determine whether expression (mRNA and protein) differences in voided urine cells are also exhibited in biopsied bladder mucosa. The investigator will use targeted assays to confirm similar methylation profiles and gene expression in voided cells and bladder biopsies. The investigator will also compare protein expression of candidate loci such as EXOC6, ZFC3H1, RPS6KA2, and SPON2 proteins, if confirmed in other Aims, between cohorts. When the proposed studies have been completed, it is the expectation that the investigator will have functionally characterized the methylation changes that the investigator preliminarily identified in IR associated OAB.

ELIGIBILITY:
Inclusion criteria:

* Women over the age of 18.
* Urgency incontinence (at least 3 times per week) for > 3months
* History of elevated A1C or Type II diabetes (UUI+IR and IR only groups)
* Non-pregnant
* At least 6 months since most recent childbirth

Exclusion criteria:

* Active pregnancy, or within 6 months of childbirth
* Breastfeeding
* Proteinuria (defined as >1+ protein on urine dipstick in the absence of infection)
* Gross hematuria (in the absence of UTI)
* Type I diabetes mellitus
* Type II diabetes with chronic renal impairment (Cr >1.5)
* Chronic renal disease (includes vasculitis, focal segmental glomerulosclerosis, lupus nephritis, polycystic kidney disease, nephropathy)
* Receiving chemotherapy or radiation for malignancy
* Taking one of the following drugs that influence DNA methylation: hydralazine, procainamide, methotrexate, valproic acid, tamoxifen, raloxifene, letrozole, anastrozole (Arimidex), or exemestane (Aromasin)
* Any history of urinary tract malignancy (bladder, urethra, ureter, kidney)
* Intradetrusor Botox injection within the prior 12 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit of a total of 450 women from three groups (at least 130 women in each cohort: 1) OAB and IR; 2) IR only; and 3) OAB only) to provide limited clinical information, blood, and urine samples. A subset of these participants (20 from each group, or 60 total) will be further recruited to provide non-muscle invasive (urothelium only) bladder biopsies. Women will be recruited through advertising and from clinical sites at Duke University Health System.
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Proportions of differentially methylated CpG sites between cohorts, from Illumina EPIC chip | 2 years
  Extract DNA from voided urine cells and compare human DNA using Illumina EPIC Methylation Chip to assess methylation of different sites across the genome

SECONDARY OUTCOMES:
Compare methylation between DNA extracted from voided urine cells and bladder urothelial biopsies | 2 years
  DNA will be extracted from voided urine cells and from urothelial biopsies in the same patients. Targeted methylation assays will be used to compare methylation sites between sample types
Gene expression (from RNA-sequencing) | 2 Years
  Compare mRNA recovered from bladder biopsies between women in 3 cohorts (Urgency incontinence only, insulin resistance only, urgency incontinence with insulin resistance)
Gene expression (from PCR) | 2 Years
  Compare expression of candidate genes between cohorts by using polymerase chain reaction (PCR) and extracted RNA

CONTACTS AND LOCATIONS:
Overall Officials: Nazema Y Siddiqui, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No